CLINICAL TRIAL: NCT04814173
Title: Evaluation of the Efficacy of One-jaw Versus Tow-jaw Mechanics for Mini-implants Anchored Total-maxillary-arch-distalization in the Treatment of Class II Division 1 Malocclusion A Randomized Controlled Trial
Brief Title: The Efficacy of Tow Mechanics for Total-maxillary-arch-distalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hama University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2021-03-14; First posted 2021-03-24 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2021-03

CONDITIONS: Malocclusion; Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion; Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One jaw mechanic (Experimental): Mini-implants anchored total-maxillary-arch-distalization using a one-jaw mechanic (mini-implants in the maxillary arch).
  Interventions: Other: One-jaw mechanic total maxillary arch distalization
- Two-jaw mechanic (Experimental): Mini-implants anchored total-maxillary-arch-distalization using a two-jaw mechanic (mini-implants in the mandibular arch with class II elastics).
  Interventions: Other: Two-jaw mechanic total maxillary arch distalization
- Traditional treatment (Experimental): traditional en-mass retraction with first premolars extraction with mini-implants in the maxillary arch.
  Interventions: Other: en-mass retraction

INTERVENTIONS:
Other: One-jaw mechanic total maxillary arch distalization — A group of patients in which participants will be undergo to the one-jaw mechanic for mini-implants anchored total-maxillary-arch-distalization (the mini-implants will be inserted in the maxillary arch between the roots of 2nd premolar and 1st molar and closer to the molar, then a force of 250 g will be applied from the TAD to a hook lateral to the laterals).
  Arms: One jaw mechanic
Other: Two-jaw mechanic total maxillary arch distalization — A group of patients in which participants will be undergo to the tow-jaw mechanic for mini-implants anchored total-maxillary-arch-distalization (the mini-implants will be inserted in the mandibular arch between the 2nd premolar and 1st molar, then, a class II elastics 3/16 and 6.5oz will be use from the TAD to the hook of canines brackets).
  Arms: Two-jaw mechanic
Other: en-mass retraction — A group of patients in which participants will be undergo to the en-mass retraction with first premolars extraction with mini-implants in the maxillary arch inserted between the 2nd premolar and 1st molar, then a force of 250 g will be applied from the TAD to a hook lateral to the laterals .
  Arms: Traditional treatment

SUMMARY:
Patients with class II division 1 malocclusion who have increased overjet will be treated in this study. The efficacy of one-jaw and tow-jaw mechanics for mini-implants anchored total-maxillary-arch-distalization in the treatment of class II division 1 malocclusion will be assessed. The skeletal, dental and soft tissues changes resulted by these tow interventions will be studied. As well as, the pain levels, oral-health related quality of life during all stages of the treatment and the smile components will be explored and compared with the traditional treatment results of this type of malocclusion (en-mass retraction with first premolars extraction).

There are three groups :

1. a group of patients in which participants will be undergo to the one-jaw mechanic for mini-implants anchored total-maxillary-arch-distalization (mini-implants in the maxillary arch).
2. a group of patients in which participants will be undergo to the tow-jaw mechanic for mini-implants anchored total-maxillary-arch-distalization (mini-implants in the mandibular arch with class II elastics).
3. a group of patients in which participants will be undergo to the en-mass retraction with first premolars extraction with mini-implants in the maxillary arch.

DETAILED DESCRIPTION:
The number of adults seeking active orthodontic treatment has been increasing over the past several decades. Older patients tend to show a greater demand for esthetic considerations during and after active treatment. Also, the preservation of existing dentoalveolar structures becomes a more critical issue in their treatment, and this mandates vigilant monitoring of the periodontal and occlusal statuses throughout the course of tooth movement.

Nowadays, the tendency towards choosing nonextraction approaches has been increasing because of the availability of effective and minimally invasive treatment modalities. Several strategies have been introduced to address the arch length discrepancy by gaining space through enamel stripping, arch expansion, and distalization of dentition. Moreover, the introduction of temporary anchorage devices (TADs) has enhanced the efficiency of nonextraction therapies via improved anchorage management.

The total-maxillary-arch-distalization is a treatment modality respect the principle of structures preservation and the esthetic demands of patients.

Most of the published literature were case reports or retrospective studies so, there is a high need for a randomized controlled trial to assess some of these suggested approaches.

The current study will have three parallel arms as following:

1. Group 1: a group of patients in which participants will be undergo to the one-jaw mechanic for mini-implants anchored total-maxillary-arch-distalization (the mini-implants will be inserted in the maxillary arch between the roots of 2nd premolar and 1st molar and closer to the molar, then a force of 250 g will be applied from the TAD to a hook lateral to the laterals).
2. a group of patients in which participants will be undergo to the tow-jaw mechanic for mini-implants anchored total-maxillary-arch-distalization (the mini-implants will be inserted in the mandibular arch between the 2nd premolar and 1st molar, then, a class II elastics 3/16 and 6.5oz will be use from the TAD to the hook of canines brackets).
3. a group of patients in which participants will be undergo to the en-mass retraction with first premolars extraction with mini-implants in the maxillary arch inserted between the 2nd premolar and 1st molar, then a force of 250 g will be applied from the TAD to a hook lateral to the laterals .

Prior to enrollment of each subject into the study, they will be examined completely to determine the orthodontic treatment plan. The operator will inform them about the aim of the study and ask them to provide a written informed consent.

A fixed orthodontic appliance will be bonded ( MBT 0.022 inch prescription), the active distalization or retraction will start when the rectangular stainless steel archwires (0.019" × 0.025").

The end of the treatment will be determined clinically when a class I canine relationship achieved with a good incisor relationship obtained.

Dental casts will be used for the quantification of the anteroposterior movement of the anterior teeth and the first molars before the beginning of the treatment and when a class I canine relationship achieved with a good incisor relationship obtained.

Cephalograms will be taken 3 times: the first before the beginning treatment for diagnosis purpose, the second: after the completion of leveling and alignment stage, the third: when a class I canine relationship achieved with a good incisor relationship obtained.

Smile photographs will be taken in 2 times: the first before the beginning of the treatment, the second: after the treatment

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with permanent occlusion at age 18-30 years.
* Comprehensive medical and dental history ruling out any systemic disease
* Not under any systemic medication.
* No previous orthodontic treatment
* Patients with satisfactory periodontal health and Good oral hygiene
* Need to orthodontic treatment with fixed appliances
* No congenitally missing teeth except third molars in the maxillary arch
* Mild or no anterior crowding in maxillary arch.
* Patients with class Ⅱ division 1 (ANB angle ≤7 degrees) with severe overjet (5-9 mm)
* Maximum retraction of the anterior teeth was desired.

Exclusion Criteria:

* Patients with previous orthodontic treatment.
* Patients with severe skeletal dysplasia in all three dimensions.
* Patients suffer from systemic diseases or syndromes
* Patients on medication for systemic disorders, pregnancy or steroid therapy.
* Patients showing any signs of active periodontal disease
* Patients with severe crowding (≥ 3.5 mm) in maxillary arch
* Patients with missing or extracted teeth in maxillary arch except third molar.

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Duration of the treatment | duration (in months) between T0: the beginning of active treatment, T1: when a normal overjet and canines class I relationships achieved. (expected to be within 6 months in the exp. groups and 8 months in the control group)
  Assessment will be performed by calculating the months required to achieve a normal overjet and canines class I relationships through clinical examination
Change in the Incisors' positions | : T0: 1 day before the beginning of active treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6 months in the exp. groups and 8 months in the control group
  Amount of distance being traveled by the retracted anterior teeth is going to be measured on study models taken when a normal overjet and canines class I relationships will be achieved.
Change in Molars' positions | : T0: 1 day before the beginning of active treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6 months in the exp. groups and 8 months in the control group
  Amount of distance being traveled by the first molars and is going to be measured on study models taken when a normal overjet and canines class I relationships will be achieved.
Change in the SNA angle | : T0: 1 day before the beginning of active treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6 months in the exp. groups and 8 months in the control group
  This angle represents the position of the upper jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the SNB angle | : T0: 1 day before the beginning of active treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6 months in the exp. groups and 8 months in the control group
  This angle the represents the position of the lower jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the ANB angle | : T0: 1 day before the beginning of active treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6 months in the exp. groups and 8 months in the control group
  This angle the represents the spatial relationship between the upper and lower jaws in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the SN.GoMe angle | : T0: 1 day before the beginning of active treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6 months in the exp. groups and 8 months in the control group
  This angle the represents the amount of backward rotation of the lower jaw in the cephalometric analysis. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the MM angle | : T0: 1 day before the beginning of active treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6 months in the exp. groups and 8 months in the control group
  This angle the represents the amount of vertical divergence between the upper and lower jaws in the cephalometric analysis. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the nasolabial angle | : T0: 1 day before the beginning of active treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6 months in the exp. groups and 8 months in the control group
  This angle the represents the relationship of the upper lip with the nose in the cephalometric analysis. Lateral cephalograms will be taken and this angle is going to be measured in degrees.

SECONDARY OUTCOMES:
Change in the levels of spontaneous and chewing pain | Levels of pain will be assessed at : immediately after the begging of the distalization or retraction (T1), 6 hours (T2) , 24 hours (T3) , 48 hours (T4), 1 week (T5) and 24 hours of each force activation.
  Assessment will be performed using questionnaires via visual analog scales (VAS).0 indicated 'no pain' and 10 indicated the 'extreme level of pain' perception.
Change in the smile components | T0: 1 day before the beginning of the treatment . T1: at the end of the treatment (expected to be within 6 months in the exp. groups and 8 months in the control group)
  The smile photographs will be analyzed using a Smile Mesh which assess the following components: Maximum incisor exposure, Upper lip drape, Lower lip to maxillary incisor, Interlabial gap, Visible posterior tooth width, Smile width, Smile index, Commissure corridor left, Commissure corridor right, Buccal corridor left, Buccal corridor right, Buccal corridor ratio, Upper lip thickness andLower lip thickness. All these components will be measured with millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Syrian Arab Republic -Department of Orhodontic, University of Hama, Hama, Hama City, Syria

REFERENCES:
- [Background] Choi YJ, Lee JS, Cha JY, Park YC. Total distalization of the maxillary arch in a patient with skeletal Class II malocclusion. Am J Orthod Dentofacial Orthop. 2011 Jun;139(6):823-33. doi: 10.1016/j.ajodo.2009.07.026. PMID 21640890
- [Background] Bechtold TE, Kim JW, Choi TH, Park YC, Lee KJ. Distalization pattern of the maxillary arch depending on the number of orthodontic miniscrews. Angle Orthod. 2013 Mar;83(2):266-73. doi: 10.2319/032212-123.1. Epub 2012 Sep 12. PMID 22970751
- [Background] Chen G, Teng F, Xu TM. Distalization of the maxillary and mandibular dentitions with miniscrew anchorage in a patient with moderate Class I bimaxillary dentoalveolar protrusion. Am J Orthod Dentofacial Orthop. 2016 Mar;149(3):401-10. doi: 10.1016/j.ajodo.2015.04.041. PMID 26926028
- [Background] Park CO, Sa'aed NL, Bayome M, Park JH, Kook YA, Park YS, Han SH. Comparison of treatment effects between the modified C-palatal plate and cervical pull headgear for total arch distalization in adults. Korean J Orthod. 2017 Nov;47(6):375-383. doi: 10.4041/kjod.2017.47.6.375. Epub 2017 Sep 29. PMID 29090125
- [Background] Jo SY, Bayome M, Park J, Lim HJ, Kook YA, Han SH. Comparison of treatment effects between four premolar extraction and total arch distalization using the modified C-palatal plate. Korean J Orthod. 2018 Jul;48(4):224-235. doi: 10.4041/kjod.2018.48.4.224. Epub 2018 Jul 6. PMID 30003056
- [Background] Shoaib AM, Park JH, Bayome M, Abbas NH, Alfaifi M, Kook YA. Treatment stability after total maxillary arch distalization with modified C-palatal plates in adults. Am J Orthod Dentofacial Orthop. 2019 Dec;156(6):832-839. doi: 10.1016/j.ajodo.2019.01.021. PMID 31784017